CLINICAL TRIAL: NCT01355796
Title: Randomized Cross Over Study of Inhaled Hypertonic Xylitol Versus Hypertonic Saline in Stable Subjects With Cystic Fibrosis
Brief Title: Inhaled Xylitol Versus Saline in Stable Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joseph Zabner (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); Northwestern University (Other)
Responsible Party: Sponsor-Investigator, Joseph Zabner, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201209728
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Xylitol; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aerosolized Hypertonic xyltiol (Experimental): Aerosolized xylitol (5 ml) twice daily for 14 days
  Interventions: Drug: Xylitol; Drug: Hypertonic saline
- Hypertonic saline (Active Comparator): Aerosolized 7% hypertonic saline (4 ml) twice daily for 14 days
  Interventions: Drug: Xylitol; Drug: Hypertonic saline

INTERVENTIONS:
Drug: Xylitol — Aerosolized 15% xylitol, 5 ml twice a day for 2 weeks
  Other Names: Xylo-pentane-1, 2, 3, 4, 5-pentol
Drug: Hypertonic saline — 4 ml of 7 % saline aerosolized twice a day for 2 weeks
  Other Names: 7% NaCl

SUMMARY:
Cystic fibrosis (CF) lung disease is characterized by chronic bacterial colonization and recurrent infection of the airways. Lowering the airway surface liquid (ASL) salt concentration has been shown to increase activity of salt sensitive antimicrobial peptides.

Xylitol is a 5-carbon sugar that can lower the ASL salt concentration, thus enhancing innate immunity.In this study, the investigators plan to study the safety and efficacy of 2 weeks of inhaled xylitol compared to 2 weeks of hypertonic saline in a randomized crossover design in stable subjects with cystic fibrosis

DETAILED DESCRIPTION:
Cystic fibrosis (CF) lung disease is characterized by chronic bacterial colonization and recurrent infection of the airways. Disruption of the cystic fibrosis transmembrane conductance regulator chloride channels in subjects with CF results in altered fluid and electrolyte transport across the airway epithelium thereby initiating infections.

These infections eventually destroy the lungs and contribute to significant morbidity and mortality in patients with CF. It is well known that antibacterial activity of innate immune mediators such as lysozyme and beta defensins in human airway surface liquid (ASL) is salt-sensitive; an increase in salt concentration inhibits their activity.

Conversely, their activity is increased by low ionic strength. Lowering the ASL salt concentration and increasing the ASL volume might therefore potentiate innate immunity and therefore decrease or prevent airway infections in subjects with CF.

Xylitol, a five-carbon sugar with low transepithelial permeability, which is poorly metabolized by bacteria can lower the salt concentration of both cystic fibrosis (CF) and non-CF epithelia in vitro. Xylitol is an artificial sweetener that has been successfully used in chewing gums to prevent dental caries; it has been used as an oral sugar substitute without significant adverse effects. It has also been shown to decrease the incidence of acute otitis media by 20-40%; nasal application to normal human subjects was found to decrease colonization with coagulase negative staphylococcus. The investigators found that aerosolized iso-osmolar xylitol was safe in mice, healthy volunteers and stable subjects with CF when administered over a single day. In a recent study, the investigators observed that single doses of 10% followed by 15% xylitol was well tolerated by subjects with cystic fibrosis who were stable.

In this study, the investigators plan to study the safety and efficacy of 2 weeks of inhaled xylitol compared to 2 weeks of hypertonic saline in a randomized crossover design in stable subjects with cystic fibrosis

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CF (medical record evidence of 2 identified CFTR(Cystic fibrosis transmembrane conductance regulator) mutations or a positive sweat chloride test or nasal voltage difference, and 1 or more clinical findings of CF)
* Age 16 or greater
* FEV1>30% predicted
* Oxygen saturation > or equal too 90% on room air
* Clinically stable, without evidence of pulmona4ry exacerbation for at least 2 weeks prior to screening (defined as use of oral or intravenous antibiotics for cystic fibrosis exacerbation)
* Use of effective contraception in women
* Ability to provide written informed consent and assent
* Successful completion of the trial doses of study drugs

Exclusion Criteria:

* Pregnancy
* Hemoptysis more than 100 mL within the last 30 days
* Change in chronic medication within the last 30 days
* History of elevated serum creatinine (> than or equal to 2 mg/dl) within 30 days or at screening
* History of lung and other solid organ transplantation
* Wait-listed for lung or other solid organ transplant
* Known intolerance to inhaled hypertonic saline

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zabner, MD, Principal Investigator — University of Iowa; Lakshmi Durairaj, MD, Study Director — University of Iowa
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois

REFERENCES:
- [Background] Rowe SM, Miller S, Sorscher EJ. Cystic fibrosis. N Engl J Med. 2005 May 12;352(19):1992-2001. doi: 10.1056/NEJMra043184. No abstract available. PMID 15888700
- [Background] Zabner J, Smith JJ, Karp PH, Widdicombe JH, Welsh MJ. Loss of CFTR chloride channels alters salt absorption by cystic fibrosis airway epithelia in vitro. Mol Cell. 1998 Sep;2(3):397-403. doi: 10.1016/s1097-2765(00)80284-1. PMID 9774978
- [Background] Goldman MJ, Anderson GM, Stolzenberg ED, Kari UP, Zasloff M, Wilson JM. Human beta-defensin-1 is a salt-sensitive antibiotic in lung that is inactivated in cystic fibrosis. Cell. 1997 Feb 21;88(4):553-60. doi: 10.1016/s0092-8674(00)81895-4. PMID 9038346
- [Background] Bals R, Wang X, Wu Z, Freeman T, Bafna V, Zasloff M, Wilson JM. Human beta-defensin 2 is a salt-sensitive peptide antibiotic expressed in human lung. J Clin Invest. 1998 Sep 1;102(5):874-80. doi: 10.1172/JCI2410. PMID 9727055
- [Background] Travis SM, Conway BA, Zabner J, Smith JJ, Anderson NN, Singh PK, Greenberg EP, Welsh MJ. Activity of abundant antimicrobials of the human airway. Am J Respir Cell Mol Biol. 1999 May;20(5):872-9. doi: 10.1165/ajrcmb.20.5.3572. PMID 10226057
- [Background] Makinen KK, Bennett CA, Hujoel PP, Isokangas PJ, Isotupa KP, Pape HR Jr, Makinen PL. Xylitol chewing gums and caries rates: a 40-month cohort study. J Dent Res. 1995 Dec;74(12):1904-13. doi: 10.1177/00220345950740121501. PMID 8600188
- [Background] Soderling E, Makinen KK, Chen CY, Pape HR Jr, Loesche W, Makinen PL. Effect of sorbitol, xylitol, and xylitol/sorbitol chewing gums on dental plaque. Caries Res. 1989;23(5):378-84. doi: 10.1159/000261212. PMID 2766327
- [Background] Makinen KK. Long-term tolerance of healthy human subjects to high amounts of xylitol and fructose: general and biochemical findings. Int Z Vitam Ernahrungsforsch Beih. 1976;15:92-104. PMID 783060
- [Background] Uhari M, Kontiokari T, Koskela M, Niemela M. Xylitol chewing gum in prevention of acute otitis media: double blind randomised trial. BMJ. 1996 Nov 9;313(7066):1180-4. doi: 10.1136/bmj.313.7066.1180. PMID 8916749
- [Background] Durairaj L, Launspach J, Watt JL, Businga TR, Kline JN, Thorne PS, Zabner J. Safety assessment of inhaled xylitol in mice and healthy volunteers. Respir Res. 2004 Sep 16;5(1):13. doi: 10.1186/1465-9921-5-13. PMID 15377394
- [Background] Singh PK, Jia HP, Wiles K, Hesselberth J, Liu L, Conway BA, Greenberg EP, Valore EV, Welsh MJ, Ganz T, Tack BF, McCray PB Jr. Production of beta-defensins by human airway epithelia. Proc Natl Acad Sci U S A. 1998 Dec 8;95(25):14961-6. doi: 10.1073/pnas.95.25.14961. PMID 9843998
- [Background] Zabner J, Seiler MP, Launspach JL, Karp PH, Kearney WR, Look DC, Smith JJ, Welsh MJ. The osmolyte xylitol reduces the salt concentration of airway surface liquid and may enhance bacterial killing. Proc Natl Acad Sci U S A. 2000 Oct 10;97(21):11614-9. doi: 10.1073/pnas.97.21.11614. PMID 11027360
- [Background] Durairaj L, Launspach J, Watt JL, Mohamad Z, Kline J, Zabner J. Safety assessment of inhaled xylitol in subjects with cystic fibrosis. J Cyst Fibros. 2007 Jan;6(1):31-4. doi: 10.1016/j.jcf.2006.05.002. Epub 2006 Jun 15. PMID 16781897
- [Background] Durairaj L, Neelakantan S, Launspach J, Watt JL, Allaman MM, Kearney WR, Veng-Pedersen P, Zabner J. Bronchoscopic assessment of airway retention time of aerosolized xylitol. Respir Res. 2006 Feb 16;7(1):27. doi: 10.1186/1465-9921-7-27. PMID 16483382
- [Background] Marks JH, Hare KL, Saunders RA, Homnick DN. Pulmonary function and sputum production in patients with cystic fibrosis: a pilot study comparing the PercussiveTech HF device and standard chest physiotherapy. Chest. 2004 Apr;125(4):1507-11. doi: 10.1378/chest.125.4.1507. PMID 15078765

RESULTS

PARTICIPANT FLOW:
Groups:
- Xylitol First Then Saline: Drug
  Xylitol: Aerosolized 15% xylitol, 5 ml twice a day for 14 days Xylo-pentane-1,2,3,4 5-pentol: 5 ml of 15 % aerosolized 2 times per day
  Saline:
  Hypersal: Hypertonic saline 7%, 4 ml twice a day for 14 days
- Saline First and Then Xylitol: Aerosolized 7% hypertonic saline (4 ml) twice daily for 14 days
  Xylitol: Aerosolized 15% xylitol, 5 ml twice a day for 2 weeks
  Xylo-pentane-1,2,3,4 5-pentol: 5 ml of 15 % aerosolized 2 times per day
Period: Overall Study
Arm/Group | Xylitol First Then Saline | Saline First and Then Xylitol
Started | 15 | 15
First Intervention for 14 Days | 15 | 15
Washout Period for 7 Days | 15 | 15
Second Intervention for 14 Days | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Baseline characteristics of the entire study cohort
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 26
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 30
FEV1 [Mean (Inter-Quartile Range); unit: % of predicted] | 71 [64 to 78]

OUTCOME MEASURES:

1. Primary Outcome: Change in FEV1 % Predicted From Baseline
Description: Change from baseline in FEV1(maximal amount of air you can forcefully exhale in one second) % predicted
Time Frame: Baseline and 14 days
Measure: Mean (95% Confidence Interval); unit: percentage of predicted
Groups:
- Xylitol: Drug
  Aerosolized xylitol (5 ml) twice daily for 14 days
  Xylitol: Aerosolized 15% xylitol, 5 ml twice a day for 2 weeks, Xylo-pentane-1,2,3,4 5-pentol: 5 ml of 15 % aerosolized 2 times per day
- Saline: Hypersal, 7%, 4 ml BID
Arm/Group | Xylitol | Saline
Number analyzed (Participants) | 30 | 30
percentage of predicted | -0.1 [-2.4 to 2.2] | 1.4 [-0.92 to 3.7]
Statistical Analysis 1: Comparison: Xylitol vs Saline; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = 1.49, 95% CI 2-sided [-1.76 to 4.75], Standard Error of Mean 1.66

2. Secondary Outcome: Sputum Density
Description: Difference from baseline in density of Pseudomonas aeruginosa colonization per gram of sputum,
Time Frame: baseline and 14 days
Population: 27 out of 30 subjects were able to give sputum on day 14 and only those subjects are included in this analysis
Measure: Mean (95% Confidence Interval); unit: Log colony forming units
Arm/Group | Xylitol | Saline
Number analyzed (Participants) | 27 | 27
Log colony forming units | -1.98 [-4.07 to 0.11] | 0.93 [-0.90 to 2.77]

ADVERSE EVENTS:
Time Frame: Average of 21 days (14 days of study drug use and 7 days after the last study drug use.
Groups:
- Aerosolized Hypertonic Xyltiol: Drug
  Aerosolized xylitol (5 ml) twice daily for 14 days
  Xylitol: Aerosolized 15% xylitol, 5 ml twice a day for 2 weeks
  Xylo-pentane-1,2,3,4 5-pentol: 5 ml of 15 % aerosolized 2 times per day
- Hypertonic Saline: Aerosolized 7% hypertonic saline (4 ml) twice daily for 14 days
  Xylitol: Aerosolized 15% xylitol, 5 ml twice a day for 2 weeks
  Xylo-pentane-1,2,3,4 5-pentol: 5 ml of 15 % aerosolized 2 times per day
Arm/Group | Aerosolized Hypertonic Xyltiol | Hypertonic Saline
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/30
Other Adverse Events (participants affected / at risk) | 1/30 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerosolized Hypertonic Xyltiol (N=30) | Hypertonic Saline (N=30)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aerosolized Hypertonic Xyltiol (N=30) | Hypertonic Saline (N=30)
headache (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No